CLINICAL TRIAL: NCT00103831
Title: Phase I Alimta Combination With BMS-275183 (Oral Taxane)
Brief Title: Oral Taxane in Combination With Pemetrexed (Alimta) in Patients With Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: CA165-021
Record Dates: First submitted 2005-02-15; First posted 2005-02-16 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC - non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — taxane

INTERVENTIONS:
Drug: Oral Taxane

SUMMARY:
A phase I-II dose ranging study of BMS-275183 (oral taxane) in combination with pemetrexed (Alimta) in patients with recurrent Non-Small Cell Lung Cancer (NSCLC). The safety and efficacy of this combination will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic pretreated NSCLC
* Measurable disease
* Adequate hematologic, hepatic and renal functions.
* ECOG Performance Status 0-2

Exclusion Criteria:

* Inability to swallow capsules
* Recent significant cardiovascular disease
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Local Institution, Denver, Colorado
  - Local Institution, Rochester, Minnesota
- Local Institution, Toronto, Ontario, Canada